CLINICAL TRIAL: NCT01952652
Title: Comparison of Post-operative Analgesic Effects of Naproxen Sodium and Naproxen Sodium-codeine Phosphate Administered Preemptively for Arthroscopic Meniscus Surgery
Brief Title: Naproxen Codeine in Arthroscopic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, CAGLA BALI,MD, MD,Anesthesiology and Reanimation, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KA12/268
Record Dates: First submitted 2013-09-20; First posted 2013-09-30 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Arthroscopic Meniscus Surgery
Keywords: Naproxen-codeine; preemptive analgesia; day case surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Naproxen sodium (Group N) (Active Comparator): Group N received naproxen sodium 550 mg 60 minutes before surgery.
  Interventions: Drug: Group N:Naproxen sodium
- Group Naproxen sodium codeine phosphate (Group NC) (Active Comparator): Group NC received naproxen sodium 550 mg+30 mg codeine 60 minutes before surgery.
  Interventions: Drug: Group NC :naproxen sodium codeine phosphate

INTERVENTIONS:
Drug: Group N:Naproxen sodium — drug will be given 60 minutes before surgery
  Other Names: Apranax fort tb, Abdi Ibrahim Ilaç,Turkiye
  Arms: Group Naproxen sodium (Group N)
Drug: Group NC :naproxen sodium codeine phosphate — drug will be given 60 minutes before surgery
  Other Names: Apranax plus tb, Abdi Ibrahim Ilac, Turkey
  Arms: Group Naproxen sodium codeine phosphate (Group NC)

SUMMARY:
In this study, the aim is to compare the efficacy of single dose naproxen sodium and combination of naproxen sodium-codeine phosphate on post-operative pain in adult patients undergoing arthroscopic menisectomy.Pre-emptive oral naproxen-codeine may be safely and more advantageous than naproxen alone.

DETAILED DESCRIPTION:
Patients receiving preemptive oral naproxen sodium (Group N) or naproxen sodium-codeine phosphate (Group NC) were assigned in 2 groups.Preoperatively, drugs were given orally by a nurse unaware of the study to both groups within 60 minutes before surgery. Hemodynamic datas, possible side effects, pain and sedation levels of patients were recorded. Patient's pain and sedation levels were statistically assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing arthroscopic meniscectomy were included in the study.

Exclusion Criteria:

* ≤ 18 years of age
* hypersensitivity to non-steroidal anti-inflammatory drugs and codeine,
* history of peptic ulcer, gastritis, upper gastrointestinal bleeding
* coagulation disorder
* serious hepatic and renal impairment
* pregnancy
* long-term NSAID and opioid use

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Pain scores as measured by Visual Analogue Scale were significantly lower in Group Naproxen codeine (group NC) at all time points compared to Group Naproxen (group N) in 61 patients who underwent arthroscopic meniscus surgery. | postoperative 18 hours
  patients will be followed postoperatively 18 hours for pain levels

CONTACTS AND LOCATIONS:
Overall Officials: Anis Aribogan, Prof.,MD, Study Director — Baskent University School of Medicine
Locations (1):
- Baskent University School of Medicine Adana Teaching and Research Hospital, Adana, Turkey (Türkiye)